CLINICAL TRIAL: NCT04671121
Title: An Analysis of Cerebral Oximetry After Low Pressure Compared With Standard Pressure Pneumoperitoneum in Patients Undergoing Laparoscopic Nephrectomy: A Prospective Randomized Parallel-Group Study
Brief Title: Pneumoperitoneum and Cerebral Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cengiz KAYA, AssociateProfessor, MD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B.30.2.ODM.0.20.08/1725
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Laparoscopic Nephrectomy; Cerebral Oxygen Saturation
Keywords: Pneumoperitoneum; Spectroscopy; Near-infrared; Oximetry; Brain; Nephrectomy; Surgery; Laparoscopic
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: The patients were randomly classified into 2 groups. The patients given the low-pressure pneumoperitoneum (8 mmHg) treatment were called Group LP (n = 30), and the patients given the standard pressure treatment (14 mmHg) were called Group SP (n = 30). Each patient and the anesthesiologist responsible for that patient's anesthesia management were blinded to the group assignments.
Who Masked: Participant, Care Provider
Masking Description: Patients were randomly classified into 2 groups using opaque sealed envelopes. Randomization was performed using a computer-generated random number list, and a statement indicating the patient's group was placed in a closed envelope numbered according to the result. Each patient was asked to choose an envelope, and the patients were assigned to the study according to the group written in the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup LP (n = 31) (Active Comparator): CO2 insufflation pressure was kept at 8 mmHg throughout the surgery.
  Interventions: Procedure: Low pressure pneumoperitoneum
- Grup SP (n = 31) (Active Comparator): CO2 insufflation pressure was kept at 14 mmHg throughout the surgery.
  Interventions: Procedure: Standart pressure pneumoperitoneum

INTERVENTIONS:
Procedure: Standart pressure pneumoperitoneum — CO2 insufflation pressure was kept at 14 mmHg throughout the surgery.
  Arms: Grup SP (n = 31)
Procedure: Low pressure pneumoperitoneum — CO2 insufflation pressure was kept at 8 mmHg throughout the surgery.
  Arms: Grup LP (n = 31)

SUMMARY:
In this study, the changes in cerebral oxygen saturation due to low and high pressure pneumoperitoneum implementation were measured in patients who underwent laparoscopic nephrectomy. This prospective, double-blind study included 62 American Society of Anesthesiologists (ASA) PS class I-III patients aged 18-65 years who underwent laparoscopic nephrectomy (simple, partial, or radical). Patients were randomly classified into 2 groups: Group LP (n = 31) included patients who were treated with low pressure pneumoperitoneum (8 mmHg) and Group SP (n = 31) included patients who were treated with standard pressure (14 mmHg). A standard anesthesia protocol was used in both groups. Bilateral rSO2 values were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient went to the recovery unit. Data for mean arterial pressure (MAP), peak heart rate (HR), peripheral oxgen saturation (SpO2), and end-tidal carbon dioxide (ETCO2) were also recorded at the same time intervals. Arterial blood gas was analyzed in the 5th minute after induction (t1) while the patient was in the supine position, in the 5th and 30th minutes after insufflation (t2, t3) while the patient was in the lateral semi-oblique position, and again 10 minutes after desufflation (t4) while the patient was in the supine position. Patient demographic data, duration of anesthesia, duration of surgery, lateral position time, pneumoperitoneum time, and recovery time were also recorded. used in both groups. Bilateral rSO2 values were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient went to the recovery unit. Data for mean arterial pressure (MAP), peak heart rate (HR), SpO2, and ETCO2 were also recorded at the same time intervals. Arterial blood gas was analyzed in the 5th minute after induction (t1) while the patient was in the supine position, in the 5th and 30th minutes after insufflation (t2, t3) while the patient was in the lateral semi-oblique position, and again 10 minutes after desufflation (t4) while the patient was in the supine position. Patient demographic data, duration of anesthesia, duration of surgery, lateral position time, pneumoperitoneum time, and recovery time were also recorded.

DETAILED DESCRIPTION:
A total of 62 American Society of Anesthesiologists (ASA) PS class I-III patients between the ages of 18 and 65 years who were scheduled for elective laparoscopic nephrectomy (simple, partial, or radical) were included in the study.

A standard anesthesia protocol was used in both groups. Patients did not receive any sedative premedication. Upon entering the operating room, they underwent electrocardiogram, non-invasive blood pressure, peripheral oxygen saturation (SpO2), rSO2 (INVOS TM 5100C oximeter; Covidien), and neuromuscular monitoring (TOF-WatchTM SX; Organon, Dublin, Ireland). Subsequently, anesthesia was induced with propofol (1.5-2.5 mg/kg) and remifentanil (1 mcg/kg IV bolus for 30-60 seconds, then 0.25 mcg/kg/min), and rocuronium (1.2 mg/kg). Anesthesia was maintained with O2/Air (fraction of inspired oxygen of 0.40; inspiratory fresh gas flow of 2 L/min), sevoflurane (1 minimum alveolar concentration), and remifentanil IV infusion (0.1-0.25 mcg/kg/min). Radial arterial cannulation was also applied for arterial blood gas analysis and continuous blood pressure measurement. A mechanical ventilator (Draeger FabiusTM Plus anesthesia Workstation, Draeger Medical, Lübeck, Germany) was used at settings of tidal volume 7-8 mL/kg, inspirium/exprium expiratory ratio 1:2, and positive end-expiratory pressure of 5 cmH2O. With these settings, pre-insufflation Sp02 values were maintained at >96%, while the respiratory rate was determined with end-tidal CO2 (ETCO2) of 32-37 mmHg. These ventilator settings were maintained throughout the operation.

CO2 insufflation was performed using the closed Veress needle technique with electronic laparoflators in the patients who were placed in lateral semi-oblique (60°) and some flexion (jackknife) positions before the surgery was started. Intra-abdominal pressure was maintained at 8 mmHg in Group LS and at 14 mmHg in Group SP throughout the surgery.

During the operation, a neuromuscular blockade was achieved with rocuronium infusion (0.3-0.4 mg/kg/hour) with a post-tetanic count of zero. At the end of the case, extubation was provided by decurarizing the rocuronium with a combination of 0.02mg/kg atropine and 0.04 mg/kg neostigmine. All patients were followed up with nasopharyngeal temperature monitoring and were actively warmed using a forced-air warming system to ensure normothermia throughout the surgery. Patients were followed up in the recovery unit at the end of the surgery until their modified Aldrete score reached ≤9.

Hemodynamics The data of mean arterial pressure (MAP), peak heart rate (HR), SpO2, and ETCO2 were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient went to the recovery unit. MAP and HR values were kept at ±20% of preoperative values by changing the remifentanil infusion rate. Hypotension MAP was defined as <60 mmHg and bradycardia HR as 45 beats/minute, and these were treated with noradrenaline 4-8 mcg, atropine 0.5 mg. Patients who required noradrenaline or atropine more than twice were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic nephrectomy (simple, partial, or radical)
* The American Society of Anesthesiologists (ASA) physical status class I-III

Exclusion Criteria:

* Cerebrovascular diseases
* Neurological disorders
* Uncontrolled diabetes or hypertension
* Advanced organ failure
* Baseline peripheral oxygen saturation (SpO2) less than 96%
* Patients with hemoglobin <9 g/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Regional cerebral oxygen saturation (rSO2) | The rSO2 value changes were recorded from baseline until the patient was referred to the recovery unit, up to 160 minutes.
  The rSO2 measurements were made using the near-infrared spectroscopy (NIRS) method. For this, prior to induction, the cerebral oximetry sensor was placed at least 2 cm above the eyebrows and 3 cm from the midline in accordance with the manufacturer's instructions. Measurements were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient went to the recovery unit. Baseline values were accepted as measurements in the last 30 seconds of preoxygenation for 3 minutes with 80% oxygen before induction. Cerebral desaturation was defined as a decrease in the rSO2 value of more than 25% from the baseline value (if the baseline value is <50, the decrease should be more than 20%), with this condition lasting ≥15 seconds.
Arterial Blood Gas (ABG) analysis-pH | The pH values of the patients were recorded after anesthesia induction until 10 minutes after desufflation, up to 140 minutes.
  The pH value was measured in the 5th minute after induction (t1) while the patient was in the supine position, in the 5th and 30th minutes after insufflation (t2, t3) while the patient was in the lateral semi-oblique position, and again 10 minutes after desufflation (t4) while the patient was in the supine position.
Arterial blood gas analysis: partial pressure of oxygen (PO2) | The oxygen partial pressure values of the patients were recorded after anesthesia induction until 10 minutes after desufflation, up to 140 minutes.
  The PO2 value was measured in the 5th minute after induction (t1) while the patient was in the supine position, in the 5th and 30th minutes after insufflation (t2, t3) while the patient was in the lateral semi-oblique position, and again 10 minutes after desufflation (t4) while the patient was in the supine position.
Arterial blood gas analysis: partial pressure of carbon dioxide (PCO2) | The carbon dioxide partial pressure values of the patients were recorded after anesthesia induction until 10 minutes after desufflation, up to 140 minutes.
  The PCO2 value was measured in the 5th minute after induction (t1) while the patient was in the supine position, in the 5th and 30th minutes after insufflation (t2, t3) while the patient was in the lateral semi-oblique position, and again 10 minutes after desufflation (t4) while the patient was in the supine position.
Arterial blood gas analysis: Hemoglobin (Hg) value | The hemoglobin values of the patients were recorded after anesthesia induction until 10 minutes after desufflation, up to 140 min.
  The Hg value was measured in the 5th minute after induction (t1) while the patient was in the supine position, in the 5th and 30th minutes after insufflation (t2, t3) while the patient was in the lateral semi-oblique position, and again 10 minutes after desufflation (t4) while the patient was in the supine position.

SECONDARY OUTCOMES:
The mean arterial pressure (MAP) values | The mean arterial pressure was recorded from baseline until the patient was referred to the recovery unit, up to 160 minutes.
  The data of the mean arterial pressure were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient was referred to the recovery unit.
The heart rate (HR) values | The heart rate was recorded from baseline until the patient was referred to the recovery unit, up to 160 minutes.
  The data of heart rate were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient was referred to the recovery unit.
  The MAP and HR values were kept at ±20% of the preoperative values by changing the remifentanil infusion rate. Hypotension MAP was defined as <60 mmHg and bradycardia HR as 45 beats/minute, and were treated with noradrenaline 4-8 mcg and atropine 0.5 mg. Patients who required noradrenaline or atropine more than twice were excluded from the study.
Peripheral oxygen saturation (SPO2) values | The oxygen saturation was recorded from baseline until the patient was referred to the recovery unit, up to 160 minutes.
  The SPO2 data were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient was referred to the recovery unit.
Anesthesia time (min) | Anesthesia time was recorded during each operation.
  The duration of anesthesia was defined as the time the patient was under anesthesia.
Surgical Time (min) | Surgical time was recorded during each operation.
  Surgical time was defined as the time elapsed from the time the trocar insertion was completed until the surgery was completed and the trocars were removed.
Pneumoperitoneum Time (min) | The pneumoperitoneum time was recorded during each operation.
  This was defined as the time during which pneumoperitoneum was administered to the patient.
End-tidal carbon dioxide values (EtCO2) values | The end-tidal carbon dioxide partial pressure was recorded from baseline until the patient was referred to the recovery unit, up to 160 min
  The data for EtCO2 were recorded at baseline, at 1 minute after induction, and then every 5 minutes until the patient was referred to the recovery unit.
Lateral Semi-oblique Position Time (min) | The lateral semi-oblique position time was recorded during each operation.
  This was defined as the time the patient stayed in the lateral semi-oblique position.
Recovery Time (min) | The recovery time was recorded from the end of the surgery to extubation.
  The recovery time was defined as the time from discontinuation of sevoflurane and remifentanil to extubation at the end of the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz Kaya, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis Universitesi, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gipson CL, Johnson GA, Fisher R, Stewart A, Giles G, Johnson JO, Tobias JD. Changes in cerebral oximetry during peritoneal insufflation for laparoscopic procedures. J Minim Access Surg. 2006 Jun;2(2):67-72. doi: 10.4103/0972-9941.26651. PMID 21170237
- [Result] Ozdemir-van Brunschot DM, van Laarhoven KC, Scheffer GJ, Pouwels S, Wever KE, Warle MC. What is the evidence for the use of low-pressure pneumoperitoneum? A systematic review. Surg Endosc. 2016 May;30(5):2049-65. doi: 10.1007/s00464-015-4454-9. Epub 2015 Aug 15. PMID 26275545
- [Result] de Waal EE, de Vries JW, Kruitwagen CL, Kalkman CJ. The effects of low-pressure carbon dioxide pneumoperitoneum on cerebral oxygenation and cerebral blood volume in children. Anesth Analg. 2002 Mar;94(3):500-5; table of contents. doi: 10.1097/00000539-200203000-00005. PMID 11867365
- [Result] Tuna AT, Akkoyun I, Darcin S, Palabiyik O. Effects of carbon dioxide insufflation on regional cerebral oxygenation during laparoscopic surgery in children: a prospective study. Braz J Anesthesiol. 2016 May-Jun;66(3):249-53. doi: 10.1016/j.bjane.2014.10.004. Epub 2015 May 12. PMID 27108820
- [Result] Pelizzo G, Bernardi L, Carlini V, Pasqua N, Mencherini S, Maggio G, De Silvestri A, Bianchi L, Calcaterra V. Laparoscopy in children and its impact on brain oxygenation during routine inguinal hernia repair. J Minim Access Surg. 2017 Jan-Mar;13(1):51-56. doi: 10.4103/0972-9941.181800. PMID 27251842
- [Result] Oztan MO, Aydin G, Cigsar EB, Sutas Bozkurt P, Koyluoglu G. Effects of Carbon Dioxide Insufflation and Trendelenburg Position on Brain Oxygenation During Laparoscopy in Children. Surg Laparosc Endosc Percutan Tech. 2019 Apr;29(2):90-94. doi: 10.1097/SLE.0000000000000593. PMID 30395045
- [Result] Park EY, Koo BN, Min KT, Nam SH. The effect of pneumoperitoneum in the steep Trendelenburg position on cerebral oxygenation. Acta Anaesthesiol Scand. 2009 Aug;53(7):895-9. doi: 10.1111/j.1399-6576.2009.01991.x. Epub 2009 May 6. PMID 19426238
- [Result] Lee JR, Lee PB, Do SH, Jeon YT, Lee JM, Hwang JY, Han SH. The effect of gynaecological laparoscopic surgery on cerebral oxygenation. J Int Med Res. 2006 Sep-Oct;34(5):531-6. doi: 10.1177/147323000603400511. PMID 17133783
- [Result] Nasrallah G, Souki FG. Perianesthetic Management of Laparoscopic Kidney Surgery. Curr Urol Rep. 2018 Jan 18;19(1):1. doi: 10.1007/s11934-018-0757-4. PMID 29349580